CLINICAL TRIAL: NCT05365022
Title: Clinical and Radiological Results in Robotic Assisted Knee Prosthetic Surgery With ROSA® Knee System.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Borja Alcobía-Díaz MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Borja Alcobía-Díaz MD, PhD, MD, PhD. Clinical Professor, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/081-EC_P
Record Dates: First submitted 2022-02-25; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Knee Prosthetic Surgery; Robotic Assistance
Keywords: Knee prosthetic surgery robotic assistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Non-Robotic Assisted Knee Prosthetic Surgery (No Intervention)
- ROSA® System Robotic Assisted Knee Prosthetic Surgery (Active Comparator)
  Interventions: Device: ROSA® System Robotic Assisted Knee Prosthetic Surgery

INTERVENTIONS:
Device: ROSA® System Robotic Assisted Knee Prosthetic Surgery — Robotic Assisted Knee Prosthetic Surgery using ROSA® (Zimmer-Biomet) System
  Arms: ROSA® System Robotic Assisted Knee Prosthetic Surgery

SUMMARY:
Comparing clinical and radiological results of patients after prosthetic surgery conventionally with no robotic assistance and ROSA® Knee prosthetic surgery robotic assistance.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis requiring PS Knee Prosthesis

Exclusion Criteria:

* Not meeting Inclusion Criteria
* Requiring Constrained Prosthesis
* Metal Allergy
* Neurological disorders.
* Cognitive impairment
* Not giving consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Utility of ROSA® (Zimmer-Biomet) Robotic assisting system for knee prosthetic surgery | 6 months after surgery
  Correct lower limb mechanical alignment

SECONDARY OUTCOMES:
Mobility | 1 year after surgery
  Range of Motion in degrees
Technique reproducibility between surgeons | Intraoperative
  Reproducing mechanical alignment in degrees
Patient satisfaction | 1 year after surgery
  Patient satisfaction in a numeric scale from 1 to 10
Time to Recovery | 1 year after surgery
  Time to feel patients themselves better than presurgery in months
Time to home discharge | 1 month
  Hospital stay in days between surgery and discharging home
Pain Control | 1 year after surgery
  Pain measurement with Visual Analogue Scale (VAS)
Technique Timing at Operating Room (OR) | Intraoperative
  Timing in minutes to measure reproducibility between surgeons
Implant Stability | 1 year after surgery
  Presence of varus / valgus instability
Complications | 1 year after surgery
  Major /Minor Complications

CONTACTS AND LOCATIONS:
Overall Officials: Borja Alcobia-Díaz, MD, PhD, Study Chair — Clinical Assistant
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Email contact